CLINICAL TRIAL: NCT04547075
Title: Turkish Validity and Reliability of Lumbar Spine Surgery Expectation Survey
Brief Title: In Turkish Version Lumbar Spine Surgery Expectation Survey
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Ph.D., Kutahya Health Sciences University
Other Study IDs: KutahyaMSUspinesurgery
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Lumbar Radiculopathy; Lumbar Fracture; Patient Satisfaction; Patient Preference
Keywords: patient expectations; lumbar spine surgery; turkish version; validity and reliability
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Radiculopathy; Fractures, Bone; Patient Satisfaction; Patient Preference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Turkish validity and reliability — 1. Contact with developers and formation of steering committee
  2. Translation from English to Turkish
  3. Back translation from Turkish to English
  4. Comparison of translation
  5. Review of translated versions.
  6. Reaching consensus and development of pilot version
  7. Testing in clinical setting
  8. Revision of pilot version
  9. Testing of final version

SUMMARY:
The aim of this study was to determine the Turkish validity and reliability of Lumbar Spine Surgery Expectations Survey developed by Mancuso.

DETAILED DESCRIPTION:
Although success in lumbar spine surgeries depends on many factors, it has been reported that one of the most important of these factors is patient expectations. In order for patients and health professionals to have the same priorities and meet the same realistic goals, it is necessary to understand what patients expect. Lumbar spine surgery expectations scale was created by Mancuso et al. The aim of this study was to determine the Turkish validity and reliability of Lumbar Spine Surgery Expectations Survey developed by Mancuso.

ELIGIBILITY:
Inclusion Criteria:

* speak Turkish
* arescheduled for lumbar spine surgery by one of two participating spine surgeons

Exclusion Criteria:

* have cognitive deficits
* refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Kutahya Health Sciences University Hospital will be interviewed in person with two questionnaires.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Lumbar Spine Surgery Expectation Survey | 10 minutes
  The Survey has been described in detail previously with respect to validity, reliability, and factor analysis. The Survey addresses pain, function, work status, mental well-being, and anticipated future spine condition.It is prefaced by the question ''How much relief or improvement do you expect in the following areas as a result of the treatment for your spine?'' Response options are ''back to normal or complete improvement'' (4 points), ''not back to normal but a lot of improvement'' (3 points), ''a moderate amount of improvement'' (2 points), ''a little improvement'' (1 point), and ''I do not have this expectation or this expectation does not apply to me'' (0 points).
Quebeck Back Pain Disability Index | 10 minutes
  The Quebeck Back Pain Disability Index is a condition-specific measure of disability that was described by Kopec et al. The scale contains 20 daily activities and asks the patient to rate his or her degree of difficulty in performing each activity from 0 ("not difficult at all") to 5 ("unable to do"). The item scores were summed for a total score between 0 and 100, with higher numbers representing greater levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail SARACOGLU, Ph.D., Study Director — Kutahya Health Sciences University; Cihan Cihan, Ph.D., Principal Investigator — Kutahya Health Sciences University; Metehan YANA, Ph.D., Principal Investigator — Karabuk University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided